CLINICAL TRIAL: NCT02671942
Title: A Multicenter Randomized Double-blind Clinical Study Evaluated the Safety, Pharmacokinetic and Pharmacodynamic Characteristics of Roflumilast in COPD Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CTTQ-01459-IIA
Record Dates: First submitted 2016-01-25; First posted 2016-02-02 (Estimated); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: roflumilast
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Roflumilast

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- roflumilast:250μg (Active Comparator): Drug: Roflumilast Roflumilast tablets Roflumilast 250 μg tablets, orally, once daily for 12 weeks. Any participants not tolerating study treatment will be prematurely discontinued and will receive
  Interventions: Drug: Roflumilast
- roflumilast:375μg (Active Comparator): Drug: Roflumilast Roflumilast tablets Roflumilast 375 μg tablets, orally, once daily for 12 weeks. Any participants not tolerating study treatment will be prematurely discontinued and will receive
  Interventions: Drug: Roflumilast
- roflumilast:500μg (Active Comparator): Drug: Roflumilast Roflumilast tablets Roflumilast 500 μg tablets, orally, once daily for 12 weeks. Any participants not tolerating study treatment will be prematurely discontinued and will receive
  Interventions: Drug: Roflumilast
- placebo (Placebo Comparator): Drug: placebo placebo tablets placebo tablets, orally, once daily for 12 weeks. Any participants not tolerating study treatment will be prematurely discontinued and will receive
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Roflumilast
  Arms: roflumilast:250μg; roflumilast:375μg; roflumilast:500μg
Drug: Placebo
  Arms: placebo

SUMMARY:
To evaluate the safety and pharmacokinetics of different dose roflumilast in China COPD patient.

DETAILED DESCRIPTION:
Roflumilast is a product which has been approved for the treatment of severe chronic obstructive lung disease (COPD) and its approved dose is 500μg once daily. This study is primarily designed to see whether alternation in this dose can improve tolerability of Roflumilast in COPD patients. Therefore one in three patients will start roflumilast therapy at a lower dose of 250μg/375μg once daily, another one in three will only take the 500μg tablet every day (and one placebo every day). Furthermore, the study will evaluate the safety and pharmacokinetics of different dose roflumilast in China COPD patient.

Lastly, the study will investigate what the body does to roflumilast. Patients with a history of COPD for at least last 12 months and a former smoker or current smoker with history of at least 10 pack years will be invited to participate.

The Randomization visit is considered the Baseline visit and for participants that discontinue the Main Period and continue into the Down-Titration Period Day 1 of Down Titration is considered BaselineDT.

ELIGIBILITY:
Inclusion Criteria:

1. Is male or female and aged 40 or olderThe BMI≥ 19.0 kg/m2;
2. The patient with severe to very severe COPD as difine by the 2015 Gold strategy .(postbronchodilator ≤0.7,，and a postbronchodilator FEV1≤50% predicted);
3. Has a history of chronic obstructive pulmonary disease (COPD) (according to Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2015) for at least 12 months prior to Screening (Visit V0), At least two documented moderate or severe COPD exacerbations within 12 months prior to Screening (Visit 0);
4. Must be a former smoker (defined as smoking cessation at least one year ago) or current smoker both with a smoking history of at least 10 pack years;
5. Women of childbearing age must take reliable contraceptive measures
6. Signed informed consent

Exclusion Criteria:

1. Severe or very severe COPD exacerbations is still exist in screen visit(V0);
2. Lower respiratory tract infection not resolved 4 weeks prior to the baseline visit V0;
3. History of asthma diagnosis in patients < 40 years of age or relevant lung disease other than COPD;
4. relevant lung disease other than COPD,as: Bronchiectasis, Cystic fibrosis, capillary bronchitis, lung resection, lung cancer, interstitial lung disease and active tuberculosis
5. Current participation in a pulmonary rehabilitation program or completion of a pulmonary rehabilitation program within 3 months preceding the baseline visit V0
6. Known alpha-1-antitrypsin deficiency;
7. Clinically significant abnormal Laboratory examination,may due to one Undiagnosed disease
8. The patient with severe Mental or neurological disease;
9. Has a history with Suicidal ideation or depression;
10. Congestive heart failure New York Heart Association Functional Classification (NYHA) severity grade III-IV;
11. Used disabled combination medicine;
12. A serious autoimmune disease;
13. Liver dysfunction according to Child-Pugh B/C;
14. Serious acute Infectious diseases;
15. Has a history Malignant in the last 5 years;

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-06-13 (Actual); Study Completion 2018-06-13 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentrationafter versus drug dose | baseline to 8 weeks

SECONDARY OUTCOMES:
Percentage of Participants with Adverse Events of Interest | baseline to 12 weeks
  Adverse events of interest to evaluate tolerability are defined as diarrhea, nausea, headache, decreased appetite, insomnia and abdominal pain.
Change in Pre-bronchodilator Forced Expiratory Volume in First Second (FEV1) during the down titration period | baseline to 12 weeks
  FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation. Pulmonary function testing will be performed using spirometry prior to taking study medication

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Have no plan to make individual participant data available.